CLINICAL TRIAL: NCT05041374
Title: Evaluation of Patients With Gastrointestinal Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000247; 000247-DK
Record Dates: First submitted 2021-09-10; First posted 2021-09-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10-27

CONDITIONS: Lower GI Disease; Gastrointestinal Diseases
Keywords: Digestive System Diseases; Gastrointestinal Diseases; Small Bowel Disease; Upper GI Disease; Natural History
MeSH Terms: conditions — Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Patients with known or suspected gastrointestinal disease

SUMMARY:
Background:

Ongoing and future research projects that study gastrointestinal diseases depend on access to biological samples and clinical data. Researchers want to study people who are seen and treated for these diseases. This may help them assess and treat these diseases better in the future.

Objective:

To collect data and samples from people being seen and/or treated for gastrointestinal problems at NIH, to use in future research.

Eligibility:

Adults aged 18 and older who have known or suspected gastrointestinal disorders or need screening, treatment, or follow-up per current medical guidelines.

Design:

Participants will be screened with a physical exam. Their medical records will be reviewed.

Participants will be seen by doctors based on the ailment they have. Their condition will be treated just like it would at a doctor s office. But the data and samples collected will be used for future research.

Participants may give blood, urine, and/or stool samples.

If participants have an endoscopy or colonoscopy as part of their standard care and samples are taken, they may be asked to give their leftover samples to NIH. Or, they may be asked to have extra samples taken for NIH to use. These samples may include gastric acid and/or tissue from the lining of the stomach or intestines. If samples are not taken as part of their standard care, they may be asked to have samples taken for NIH to use.

Data will be stored at NIH. The data systems are password protected. Samples will be coded.

Participants will take part in the study for as long as they agree to be seen for their disease....

DETAILED DESCRIPTION:
Patients with suspected or established acute or chronic gastrointestinal diseases or who require clinical screening for gastrointestinal diseases are provided standard clinical care for their condition. Data and samples obtained during regular clinical care will be retained for future research in gastrointestinal diseases. Recommendations for other treatment options outside of the NIH will be discussed with study patients and may be discussed with their primary or referring physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, aged >= 18 years of age
2. Known or suspected gastrointestinal disorders or requiring clinical screening, management and/or treatment and follow-up per current American Gastroenterological Association (AGA), American Society for Gastrointestinal Endoscopy (ASGE) or the American Association for the Study of Liver Disease (AASLD).

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Significant medical illnesses that the investigators feel may interfere with potential evaluations.
2. Absence of a referring community physician who would be able to manage care outside of the NIH.
3. Any medical, psychiatric, or social conditions which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the patient.
4. Inability to provide informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected gastrointestinal disease.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
To collect data and samples during clinical evaluation, treatment and follow-up of participants for future use in studies of gastrointestinal diseases. | End of study
  Development of a data set comprised of results and observations obtained during standard clinical care of patients with known or suspected gastrointestinal disease and collection of samples to be used for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Kumar, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000247-DK.html